CLINICAL TRIAL: NCT04026152
Title: Using the Unified Protocol to Reduce Exercise Anxiety and Improve Adherence to a Resistance Training Program for People With Anxiety-Related Disorders: A Randomized Controlled Trial
Brief Title: Exercising With Anxiety: Can Cognitive Behavioural Techniques Help People With Anxiety-related Disorders Exercise More?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-048
Record Dates: First submitted 2019-07-07; First posted 2019-07-19 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2019-07

CONDITIONS: Anxiety Disorders; Posttraumatic Stress Disorder; Obsessive-Compulsive Disorder
Keywords: Anxiety-Related Disorder; Exercise; Resistance Training; Unified Protocol; Adherence; Randomized Controlled Trial; Physical Activity
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder; Motor Activity | interventions — Resistance Training; Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three conditions: resistance training plus Unified Protocol, resistance training, or waitlist. Participants will then complete their assigned condition. Participants who receive the waitlist condition will have the option to be re-randomized into one of the resistance training conditions after they have completed their last waitlist measure.
Masking Description: Participants will be aware of the three study conditions in order to provide informed consent for participation; however, they will not receive detailed information or materials about any condition until they have been assigned to it. The personal trainers who will be administering the resistance training sessions do not know about the presence of the waitlist or resistance training + Unified Protocol conditions. The therapist who is administering the Unified Protocol will be aware of all conditions. The Outcomes Assessor and Investigator will also be aware of all conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance training + Unified Protocol (Experimental): Participants randomly assigned to this condition will complete a resistance training program consisting of three weekly hour-long full body exercise sessions. Participants will also receive four weekly hour-long sessions with a therapist to learn cognitive-behavioural strategies to assist them with managing their anxiety when exercising. Participants will be supported by a personal trainer for six exercise session during their first month of training and will complete the remaining six sessions during this month independently. Participants will then continue to exercise independently following this first month of intervention. Participants will fill out weekly self-report measures (~20 minutes each time) via the internet during their first four weeks of study participation and at 1-week, 1-month, and 3-months (~20 minutes each time) follow-up after they have completed the supervised portion of this study.
  Interventions: Behavioral: Resistance training; Behavioral: Unified Protocol
- Resistance training (Active Comparator): Participants randomly assigned to this condition will complete a resistance training program consisting of three weekly hour-long full body exercise sessions. Participants will be supported by a personal trainer for six exercise session during their first month of training and will complete the remaining six sessions during this month independently. Participants will then continue to exercise independently following this first month of intervention. Participants will fill out weekly self-report measures (~20 minutes each time) via the internet during their first four weeks of study participation and at 1-week, 1-month, and 3-months (~20 minutes each time) follow-up after they have completed the supervised portion of this study.
  Interventions: Behavioral: Resistance training
- Waitlist (No Intervention): Participants randomly assigned to this condition will maintain their usual physical activity and exercise routine and not engage in any additional exercise than they were prior to the study. These participants will fill out questionnaires (~20 minutes each time) following randomization into this condition, once per week for four weeks, and at 1-week, 1-month, and 3-months (~20 minutes each time) follow-up. After completing the last follow-up, participants in the waitlist condition will be re-randomized into either the resistance training only or resistance training + Unified Protocol conditions.

INTERVENTIONS:
Behavioral: Resistance training — Following randomization, all participants assigned to receive the resistance training intervention will receive a comprehensive exercise program. The exercise program participants will be using is similar to past research using resistance training programs with people with anxiety-related disorders and has been developed and reviewed by a team of certified personal trainers, including the primary investigator. All participants assigned receive this resistance training intervention will complete a total of six sessions with a personal trainer and six session independently over four weeks to allow for a gradual, rather than abrupt, transition to fully independently completed exercise by the 4th week. After this time participants will be encouraged to exercise independently.
  Other Names: Exercise
  Arms: Resistance training; Resistance training + Unified Protocol
Behavioral: Unified Protocol — This intervention consists four weekly sessions adapted from the Unified Protocol. The first module is Psychoeducation and Motivational Interviewing. During this module, participants will develop an understanding of their own pattern of emotional responding to exercise as well as increasing participants' readiness and motivation for behaviour change.The second module is Cognitive Flexibility, during which participants will learn about how automatic negative interpretations can influence their emotional reactions and prevent them from considering alternative explanations. The third module is Countering Emotion-Driven Behaviours during which participants will identify and counter behaviours used to dampen strong emotions, particularly those associated with exercise. Lastly, module four will use Exposure to external and internal emotional triggers to increase participants' tolerance to the emotions that arise in exercise environments.
  Other Names: Cognitive-behavioural therapy
  Arms: Resistance training + Unified Protocol

SUMMARY:
Anxiety-related disorders such as panic disorder, social anxiety disorder, generalized anxiety disorder, and posttraumatic stress disorder are among the most prevalent mental health disorders affecting Canadian adults. Lack of access to evidence-based treatments prevents many people with high levels of anxiety from receiving appropriate care. Evidence shows that exercise is an alternative option for alleviating anxiety that could be appealing to individuals with high levels of anxiety who are unable, or unwilling, to access other evidence-based treatments. Unfortunately, people with high levels of anxiety tend to have a hard time using exercise independently as a strategy to manage their anxiety, in part, because many aspects of exercising can be anxiety-provoking (e.g., physical sensations produced by exercise, opportunities for evaluation by others, crowded exercise environments). Cognitive-behavioral techniques are therapeutic tools that could help these people overcome their anxiety about exercising and support them as they make positive health behavioural changes; however, however, no study to date has explored this possibility. The proposed study will use rigorous experimental techniques to determine whether an exercise-focused cognitive behavioural psychological intervention can support people with anxiety-related disorders to become more physically active and experience the reductions in anxiety that comes from making this lifestyle change.

DETAILED DESCRIPTION:
Exercise is a time- and cost-efficient alternative to other evidence-based treatments for anxiety (e.g., psychotherapy, pharmaceutical) that also is associated with physical health benefits. Exercise protocols such as resistance training (RT) are efficacious at reducing symptoms of anxiety-related disorders (ARDs); however, there are challenges associated with effectively implementing such protocols, most notably, that people with ARDs may avoid physical activity, including exercise. Emerging research suggests that people with ARDs experience exercise-specific anxiety (e.g., exercise-related worries, fear of physical sensations associated with exercise) and identify this exercise anxiety as a major contributor to their exercise avoidance. Consequently, exercise interventions for people with ARDs may need to target exercise anxiety to support long-term exercise engagement. Evidence-based cognitive-behavioural techniques (CBT), such as cognitive restructuring, and exposure, can alter maladaptive thinking and behavioural patterns associated with anxiety. Teaching people with ARDs how to apply CBT techniques to exercise anxiety could help increase and support their exercise behaviour; however, research has not been conducted to test this hypothesis. The primary purpose of this proposed randomized controlled trial (RCT) is to examine whether adding a form of CBT (i.e., the Unified Protocol) to a program for people with ARDs is associated with superior exercise engagement as compared to groups that do not receive this intervention. This proposed RCT will also evaluate potential predictors of exercise frequency for people with ARDs, such as exercise knowledge, exercise self-efficacy, and exercise motivation. A total of 90 physically inactive participants with ARDs will be randomized into a month of one of the following conditions: Unified Protocol + RT, RT, or waitlist (WL). All participants (except WL) will receive and follow a comprehensive instructional exercise program, consisting of three weekly full body RT workouts. Participants in both RT groups will also receive the guidance of a personal trainer during their first month of following this program. Participants in both RT groups will complete three exercise sessions each week for 4 weeks and these sessions will be composed of personal trainer and independent exercise. Participants in the Unified Protocol +RT condition will also receive four weekly individual CBT sessions designed to support adherence to the exercise sessions. Exercise frequency will be measured using the number of recorded exercise sessions (at least 30 minutes in length) and physical activity will be measured using the International Physical Activity Questionnaire-Short Form. Presence and severity of ARDs will be assessed using the Structured Clinical Administered Interview for the Diagnostic Statistical Manual of Mental Disorders-5 (SCID-5) as well as disorder-specific self-report measures. Exercise anxiety will also be measured using a questionnaire designed for this study. Exercise frequency, anxiety disorder-specific severity, and exercise anxiety will be measured at baseline, weekly during the first month of exercise, and at follow-up at 1-week, 1-month, and 3-months. Diagnostic status will be evaluated at baseline and at 1-week follow-up. Exercise knowledge, exercise self-efficacy, exercise motivation, and physical activity, will be measured at baseline, 1-week-, 1-month-, and 3-month follow-ups. Multilevel modelling will compare exercise frequency and anxiety symptoms, across groups, at each time point. This RCT will be the first to evaluate whether the Unified Protocol can support people with ARDs to increase their exercise engagement. If the Unified Protocol does increase engagement, the Unified Protocol could be used by researchers and clinicians alike to support individuals with ARDs interested in using exercise to manage their anxiety, but who are experiencing difficulty maintaining an exercise regime.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of specific phobia, agoraphobia, social anxiety disorder, generalized anxiety disorder, panic disorder, posttraumatic stress disorder, obsessive-compulsive disorder, other specified anxiety disorder, other specified obsessive-compulsive disorder, and other specified trauma- and stressor-related disorder.
* Reports experiencing anxiety about exercising

Exclusion Criteria:

* Current enrolment in cognitive-behaviour therapy
* Comorbid substance use disorder
* Taking benzodiazepines or antipsychotic medication
* At risk for suicide
* Engages in an average of four or more resistance training exercise sessions each month
* Completes 150 minutes of moderate intensity physical activity or 75 minutes of vigorous intensity physical activity each week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Anxiety severity (change) | There are eight time points where this measure will be taken, namely (1) baseline, (2) week 1, (3) week 2, (4) week 3, (5) week 4, (6) 1-week follow-up, (7) 1-month follow-up, and (8) 3-month follow-up
  Participants will complete one of the following empirically validated clinical symptom measures for their primary anxiety disorder to assess whether any changes occur from baseline to the last follow-up. Higher scores on these measures indicate more severe symptoms. The Severity Measure for Specific Phobia-Adult (SMSP-A), The Severity Measure for Agoraphobia-Adult (SMA-A), The Social Interaction Phobia Scale (SIPS), The Panic Disorder Severity Scale-Self Report (PDSS-SR), The Generalized Anxiety Disorder 7-item scale (GAD-7), The Obsessive-Compulsive Inventory-Revised (OCI-R), The Posttraumatic Stress Disorder Checklist for the Diagnostic Statistical Manual of Mental Disorders-5(PCL-5), and The Depression Anxiety and Stress 21-item (DASS-21). T scores based on means and standard deviations from non-clinical samples will be calculated and used for comparisons.
Anxiety diagnostic status (change) | There are two time points where this measure will be taken, namely (1) eligibility assessment and (2) 1-week follow-up. UPDATE: During the actual trial (to minimize participant burden) we only used this measure for the eligibility assessment.
  The Structured Clinician Administered Interview for the Diagnostic Statistical Manual of Mental Disorders-5, Research Version (SCID-5-RV) will be administered twice during this study to assess for determine participant eligibility for the study and to evaluate potential changes in diagnostic status following intervention. Participants that meet criteria for a primary diagnosis of specific phobia, agoraphobia, social anxiety disorder, generalized anxiety disorder, panic disorder, posttraumatic disorder, obsessive-compulsive disorder, other specified anxiety disorder, other specified obsessive-compulsive disorder, or other specified trauma-and stressor-related disorder, will be eligible to participate in this study. Diagnostic status will be reassessed at the 1-week follow-up to determine if changes in diagnostic status have occured.
Exercise frequency (change) | There are eight time points where this measure will be taken, namely (1) baseline, (2) week 1, (3) week 2, (4) week 3, (5) week 4, (6) 1-week follow-up, (7) 1-month follow-up, and (8) 3-month follow-up
  Exercise frequency will be measured using the number of 30 minute (or longer) exercise sessions completed by participants across time to determine if any changes in exercise frequency occur with study participation. The greater the scores on this measure, the more participants have been exercising. This data will be collected using participant tracking logs. Participants will complete an exercise log entry in their manual every time they exercise and these workouts will be verified using the date/time stamps collected whenever they scan their membership card at the gym in order to access it. Participants will also note any workouts that they complete outside the gym in their tracking logs. UPDATE: due to gym closures from the COVID-19 pandemic, we were unable to collect time-stamped frequency data. We used self-report exercise logs for this measure.
Exercise anxiety (change) | There are eight time points where this measure will be taken, namely (1) baseline, (2) week 1, (3) week 2, (4) week 3, (5) week 4, (6) 1-week follow-up, (7) 1-month follow-up, and (8) 3-month follow-up
  The Exercise Anxiety Questionnaire is a 16-item scale that was developed for the purpose of this study to evaluate whether any changes in exercise anxiety occur with participation in this study and whether these changes are associated with exercise behaviour. Items on this measure evaluate participants' experience with exercise anxiety and the effect that this anxiety has on their exercise behaviour. Items will be rated on a Likert Scale ranging from 0 (not at all) to 4 (agree very much). Items will be summed to generate total exercise anxiety scores where higher scores indicate greater exercise anxiety.
Physical activity (change) | There are four time points where this measure will be taken, namely (1) baseline, (2) 1-week follow-up, (3) 1-month follow-up, and (4) 3-month follow-up
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF) is the abbreviated version of a self-report tool for monitoring physical activity levels. The IPAQ-SF assesses physical activity over the last 7 days across four domains (i.e., during leisure time, domestic activities, occupation, and transportation, and with three intensities (i.e., low, moderate, and vigorous). Data collected from the IPAQ-SF can be reported as a continuous weekly total energy expenditure or metabolic equivalents (METs). This measure will be used to produce a total score of weekly METs-minutes/week across time in order to determine whether any changes in physical activity occur with participation in this study.

SECONDARY OUTCOMES:
Exercise self-efficacy (change) | There are four time points where this measure will be taken, namely (1) baseline, (2) 1-week follow-up, (3) 1-month follow-up, and (4) 3-month follow-up
  The Self-Efficacy to Regulate Exercise Scale (SES) is an 18-item exercise self-efficacy self-report measure. When completing this measure, participants are required to rate how certain they are that they would be able to perform their exercise routine regularly (three or more times per week) under situations that can make it hard to stick to an exercise routine. Participants provide rating using a Likert scale ranging from 0 (cannot do at all) to 100 (highly certain can do). Items are summed together to provide a total exercise self-efficacy score, with higher scores indicating greater self-efficacy. This measure will be administered several times during this study to determine whether any changes in exercise self-efficacy occur.
Exercise knowledge (change) | There are four time points where this measure will be taken, namely (1) baseline, (2) 1-week follow-up, (3) 1-month follow-up, and (4) 3-month follow-up. UPDATE: The data collected from this measure was not usable and we were unable to include it
  Participants' knowledge about basic fitness principles, primal movement patterns, and cardiorespiratory and muscular concepts will be evaluated using The Exercise and Physical Activity Knowledge Quiz. This measure was developed for this study and has not been empirically validated. Each question will be answered with either true or false and will be worth one point for correct scores. Scores on each question will be summed to generate a total score with higher scores indicating more exercise knowledge. This measure will be administered at several time points during this study to evaluate whether any changes in exercise knowledge have occured.
Exercise motivation (change) | There are four time points where this measure will be taken, namely (1) baseline, (2) 1-week follow-up, (3) 1-month follow-up, and (4) 3-month follow-up
  The Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2) is a 19-item self-report measure of five motivational factors for exercise rated on a Likert Scale ranging from 0 (not true for me) to 10 (very true for me). This measure is scored by calculating a mean score for each of the following factors with higher scores indicating responses more consistent with the factor, external regulation (i.e., satisfy external pressures or achieve external rewards), identification (i.e., acceptance of the value of exercise), introjection (i.e., internalization of external controls to avoid negative emotional states), intrinsic regulation (i.e., taking part in exercise for the enjoyment and satisfaction inherent in engaging in the behaviour), and amotivation (i.e., lacking intention to engage in exercise). This measure will be administered throughout this study to evaluate changes in exercise motivation.
Pandemic measures | At 1-week, 1-month, and 3-month follow-up for participants who participated during the pandemic.
  After the onset of the ongoing global coronavirus pandemic we received research ethics board approval to ask participants about the effect of the pandemic on their mental health and exercise behaviour. Qualitative responses were provided by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mason, MA, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlow DH, Allen LB, Choate ML. Toward a Unified Treatment for Emotional Disorders - Republished Article. Behav Ther. 2016 Nov;47(6):838-853. doi: 10.1016/j.beth.2016.11.005. Epub 2016 Nov 10. PMID 27993336
- [Background] Andrade LH, Alonso J, Mneimneh Z, Wells JE, Al-Hamzawi A, Borges G, Bromet E, Bruffaerts R, de Girolamo G, de Graaf R, Florescu S, Gureje O, Hinkov HR, Hu C, Huang Y, Hwang I, Jin R, Karam EG, Kovess-Masfety V, Levinson D, Matschinger H, O'Neill S, Posada-Villa J, Sagar R, Sampson NA, Sasu C, Stein DJ, Takeshima T, Viana MC, Xavier M, Kessler RC. Barriers to mental health treatment: results from the WHO World Mental Health surveys. Psychol Med. 2014 Apr;44(6):1303-17. doi: 10.1017/S0033291713001943. Epub 2013 Aug 9. PMID 23931656
- [Background] Asmundson GJ, Fetzner MG, Deboer LB, Powers MB, Otto MW, Smits JA. Let's get physical: a contemporary review of the anxiolytic effects of exercise for anxiety and its disorders. Depress Anxiety. 2013 Apr;30(4):362-73. doi: 10.1002/da.22043. Epub 2013 Jan 8. PMID 23300122
- [Background] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327
- [Background] Brown RA, Abrantes AM, Strong DR, Mancebo MC, Menard J, Rasmussen SA, Greenberg BD. A pilot study of moderate-intensity aerobic exercise for obsessive compulsive disorder. J Nerv Ment Dis. 2007 Jun;195(6):514-20. doi: 10.1097/01.nmd.0000253730.31610.6c. PMID 17568300
- [Background] Collins KA, Westra HA, Dozois DJ, Burns DD. Gaps in accessing treatment for anxiety and depression: challenges for the delivery of care. Clin Psychol Rev. 2004 Sep;24(5):583-616. doi: 10.1016/j.cpr.2004.06.001. PMID 15325746
- [Background] LeBouthillier DM, Asmundson GJG. The efficacy of aerobic exercise and resistance training as transdiagnostic interventions for anxiety-related disorders and constructs: A randomized controlled trial. J Anxiety Disord. 2017 Dec;52:43-52. doi: 10.1016/j.janxdis.2017.09.005. Epub 2017 Sep 23. PMID 29049901
- [Background] Mason, J. E., Faller, Y. N., LeBouthillier, D. M., & Asmundson, G. J. G. (2018). Exercise anxiety: A qualitative analysis of the barriers, facilitators, and psychological processes underlying exercise participation for people with anxiety-related disorders. Mental Health and Physical Activity. https://doi.org/10.1016/J.MHPA.2018.11.003